CLINICAL TRIAL: NCT01135368
Title: Safety and Efficacy of Lansoprazole in Patients With Reflux Disease. An Open, Single Arm, Long-term Study
Brief Title: Safety and Efficacy of Lansoprazole in Patients With Reflux Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGO K019; U1111-1115-1139 (Registry Identifier: WHO)
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-07

CONDITIONS: Gastroesophageal Reflux
Keywords: GERD; Gastroesophageal Reflux Disease; Drug Therapy
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Lansoprazole; helicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lansoprazole (Experimental): Lansoprazole 30 mg, capsules, orally, once daily for up to 8 weeks.
  Depending on response, dosage could then be decreased to 15 mg, once daily, or increased to 30 mg, twice daily for up to 4 years and 10 months.
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole — Lansoprazole capsules
  Other Names: Prevacid; Helicid; Zoton; Inhibitol; Agopton; AG-1749

SUMMARY:
The purpose of this study is to measure the safety, efficacy and quality of life of lansoprazole in patients with reflux disease over a five year period.

DETAILED DESCRIPTION:
Lansoprazole is currently approved in Germany for the treatment of erosive reflux esophagitis and active duodenal and gastric ulcer disease, and for long-term treatment including maintenance of healed reflux esophagitis and duodenal ulcer disease and treatment of pathological hypersecretory conditions such as Zollinger-Ellison syndrome.

This study was conducted to evaluate the safety, efficacy and quality of life of patients receiving up to five years of treatment with lansoprazole.

ELIGIBILITY:
Inclusion Criteria:

* Had Gastro Esophageal Reflux disease with or without oesophagitis.
* Had a history of heartburn at least for 5 days per week during the past 6 months or was receiving long-term treatment with a proton pump inhibitor and during two weeks (without proton pump inhibitor treatment) prior to enrolment.

Exclusion Criteria:

* History of surgery of stomach or oesophagus.
* Gastric ulcer (can be included after healing of gastric ulcer).
* Duodenal ulcer (can be included after healing of duodenal ulcer).
* Bleeding (melena, hematemesis).
* Severe concomitant disease (cancer, cardiovascular, renal, hepatic diseases).
* Barrett oesophagus with dysplasia.
* Complicated esophagitis (oesophageal strictures or ulcers).
* Treatment with proton pump inhibitor or Histamine receptor 2 (H2)antagonists within the previous two weeks.
* Pregnancy, wish to become pregnant, breast feeding.
* Treatment with non steroidal anti-inflammatory drugs, treatment with acetylsalicylic acid (aspirin) > 100 mg/day.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2002-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 38 investigative sites in Germany from 18 June 2002 to 24 September 2008.
Pre-assignment Details: Participants with a historical diagnosis of Gastro Esophageal Reflux disease (GERD) received treatment with Lansoprazole at the usual dosage.
Period: Overall Study
Arm/Group | Lansoprazole
Started | 506
Completed | 255
Not Completed | 251

BASELINE CHARACTERISTICS:
Arm/Group | Lansoprazole
Number analyzed (Participants) | 506
Age Continuous [Mean (Standard Deviation); unit: years] | 53.5 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218
  Male | 288
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 502
  Black | 2
  Oriental | 2
Height [Mean (Standard Deviation); unit: cm] | 171.1 (9.3)
Weight [Mean (Standard Deviation); unit: kg] | 82.2 (13.7)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/cm^2] | 28.09 (4.15)
Diagnosis of Reflux Disease [Number; unit: participants]
  First diagnosis | 150
  Recurrence | 356

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Reflux Disease Symptom - Heartburn
Description: Heartburn symptoms were assessed by the Investigator at Baseline and the Week 8 visit. The shift table below summarizes the individual transitions in symptom intensity (mild, moderate, severe or none) between Baseline (depicted in the columns) and Week 8 (depicted in the rows) for all patients.
Time Frame: Baseline and Week 8
Population: Intent to treat population, including all patients who received at least one dose of study medication and had a subsequent rating of the primary efficacy variable.
Measure: Number; unit: participants
Groups:
- None: Participants with no symptoms at Baseline.
- Mild: Participants with mild symptoms at Baseline.
- Moderate: Participants with moderate symptoms at Baseline.
- Severe: Participants with severe symptoms at Baseline.
Arm/Group | None | Mild | Moderate | Severe
Number analyzed (Participants) | 0 | 69 | 156 | 257
participants
  Week 8 Symptoms: None |  | 59 | 117 | 186
  Week 8 Symptoms: Mild |  | 7 | 27 | 43
  Week 8 Symptoms: Moderate |  | 0 | 4 | 12
  Week 8 Symptoms: Severe |  | 0 | 0 | 2
  Week 8 Missing data |  | 3 | 8 | 14

2. Primary Outcome: Change From Baseline in Reflux Disease Symptoms - Acid Regurgitation
Description: Acid regurgitation symptoms were assessed by the Investigator at Baseline and the Week 8 visit. The shift table below summarizes the individual transitions in symptom intensity (mild, moderate, severe or none) between Baseline (depicted in the columns) and Week 8 (depicted in the rows) for all patients.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | None | Mild | Moderate | Severe
Number analyzed (Participants) | 66 | 136 | 166 | 114
participants
  Week 8 Symptoms: None | 58 | 113 | 125 | 81
  Week 8 Symptoms: Mild | 4 | 19 | 28 | 22
  Week 8 Symptoms: Moderate | 1 | 0 | 2 | 3
  Week 8 Symptoms: Severe | 0 | 0 | 1 | 0
  Week 8 Missing data | 3 | 4 | 10 | 8

3. Primary Outcome: Change From Baseline in Reflux Disease Symptom - Difficulty Swallowing
Description: Difficulty swallowing symptoms were assessed by the Investigator at Baseline and the Week 8 visit. The shift table below summarizes the individual transitions in symptom intensity (mild, moderate, severe or none) between Baseline (depicted in the columns) and Week 8 (depicted in the rows) for all patients.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | None | Mild | Moderate | Severe
Number analyzed (Participants) | 316 | 102 | 45 | 19
participants
  Week 8 Symptoms: None | 293 | 89 | 33 | 13
  Week 8 Symptoms: Mild | 7 | 9 | 5 | 2
  Week 8 Symptoms: Moderate | 3 | 0 | 1 | 1
  Week 8 Symptoms: Severe | 0 | 0 | 1 | 1
  Week 8 Missing data | 13 | 4 | 5 | 2

4. Primary Outcome: Change From Baseline in Reflux Disease Symptom - Pain in Upper Abdomen
Description: Pain in the upper abdomen symptoms were assessed by the Investigator at Baseline and the Week 8 visit. The shift table below summarizes the individual transitions in symptom intensity (mild, moderate, severe or none) between Baseline (depicted in the columns) and Week 8 (depicted in the rows) for all patients.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | None | Mild | Moderate | Severe
Number analyzed (Participants) | 139 | 155 | 120 | 68
participants
  Week 8 Symptoms: None | 124 | 125 | 86 | 44
  Week 8 Symptoms: Mild | 9 | 19 | 21 | 10
  Week 8 Symptoms: Moderate | 0 | 4 | 2 | 8
  Week 8 Symptoms: Severe | 0 | 0 | 1 | 3
  Week 8 Missing data | 6 | 7 | 10 | 3

5. Primary Outcome: Change From Baseline in Reflux Disease Symptom - Nausea & Vomiting
Description: Nausea and vomiting symptoms were assessed by the Investigator at Baseline and the Week 8 visit. The shift table below summarizes the individual transitions in symptom intensity (mild, moderate, severe or none) between Baseline (depicted in the columns) and Week 8 (depicted in the rows) for all patients.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | None | Mild | Moderate | Severe
Number analyzed (Participants) | 330 | 98 | 36 | 18
participants
  Week 8 Symptoms: None | 303 | 78 | 25 | 13
  Week 8 Symptoms: Mild | 10 | 9 | 9 | 2
  Week 8 Symptoms: Moderate | 2 | 1 | 2 | 2
  Week 8 Symptoms: Severe | 0 | 0 | 0 | 0
  Week 8 Missing data | 15 | 10 | 0 | 1

6. Primary Outcome: Change From Baseline in Reflux Disease Symptom - Cough & Sore Throat
Description: Cough and sore throat symptoms were assessed by the Investigator at Baseline and the Week 8 visit. The shift table below summarizes the individual transitions in symptom intensity (mild, moderate, severe or none) between Baseline (depicted in the columns) and Week 8 (depicted in the rows) for all patients.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | None | Mild | Moderate | Severe
Number analyzed (Participants) | 343 | 81 | 35 | 23
participants
  Week 8 Symptoms: None | 305 | 71 | 24 | 14
  Week 8 Symptoms: Mild | 16 | 4 | 7 | 6
  Week 8 Symptoms: Moderate | 3 | 3 | 0 | 2
  Week 8 Symptoms: Severe | 0 | 0 | 0 | 0
  Week 8 Missing data | 19 | 3 | 4 | 1

7. Primary Outcome: Change From Baseline in Endoscopic Healing of Erosive Reflux Disease as Assessed by Endoscopy
Description: Los Angeles Classification is used to grade the extension of changes in the oesophagus induced by reflux disease (Grade 0: normal aspect of mucosa; Grade A: ≥1 mucosal breaks no longer than 5 mm; Grade B: ≥1 mucosal breaks >5 mm long; Grade C: mucosal breaks extending between tops of two or more mucosal folds but are <75% of the circumference; Grade D: mucosal breaks ≥75% of the circumference). Healed defined as anything less than Grade A criteria. The shift table below summarizes the individual transitions in Los Angeles classification between Baseline (table columns) and Week 8 (table rows).
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Grade 0: Participants with Grade 0 (normal aspect of mucosa) at Baseline.
- Grade A: Participants with Grade A (one or more mucosal breaks no longer than 5 mm, none of which extends between the tops of the mucosal folds) at Baseline.
- Grade B: Participants with Grade B (one or more mucosal breaks more than 5 mm long, none of which extends between the tops of two mucosal folds) at Baseline.
- Grade C: Participants with Grade C (mucosal breaks that extend between the tops of two or more mucosal folds, but which involve less than 75% of the oesophageal circumference) at Baseline.
- Grade D: Participants with Grade D (mucosal breaks which involve at least 75% of the oesophageal circumference) at Baseline.
Arm/Group | Grade 0 | Grade A | Grade B | Grade C | Grade D
Number analyzed (Participants) | 168 | 149 | 118 | 39 | 8
participants
  Week 8: Grade 0 | 38 | 97 | 79 | 17 | 4
  Week 8: Grade A | 0 | 17 | 19 | 6 | 2
  Week 8: Grade B | 0 | 0 | 3 | 1 | 1
  Week 8: Grade C | 0 | 0 | 0 | 1 | 1
  Week 8: No data | 130 | 35 | 17 | 14 | 0

8. Secondary Outcome: Change From Baseline in Enterochromaffin-like Cell Hyperplasia
Description: Enterochromaffin-like (ECL) cells were evaluated and classified by histopathological examinations as Normal, Simple (diffuse) hyperplasia, or Linear, chain producing hyperplasia.
  The shift table below summarizes the individual transitions in ECL-cell classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows) for all patients.
Time Frame: Baseline and Year 5
Population: Safety analysis set, including all participants who received any study medication. Last observation carried forward was utilized.
Measure: Number; unit: participants
Groups:
- Normal: Participants with normal ECL cell classification at Baseline.
- Simple: Participants with simple (diffuse) hyperplasia at Baseline.
- Linear: Participants with linear, chain producing hyperplasia at Baseline.
- No Data: Participants with no data at Baseline.
Arm/Group | Normal | Simple | Linear | No Data
Number analyzed (Participants) | 446 | 13 | 1 | 46
participants
  Year 5: Normal | 315 | 8 | 1 | 26
  Year 5: Simple hyperplasia | 10 | 2 | 0 | 4
  Year 5: Linear hyperplasia | 13 | 0 | 0 | 2
  Year 5: No data | 108 | 3 | 0 | 14

9. Secondary Outcome: Change From Baseline in Antrum Atrophy
Description: Atrophy was assessed by histopathological examination of cells biopsied from the antrum and classified according to the Sydney classification as mild, moderate, severe or none. The shift table below summarizes the individual transitions in atrophy classification (mild, moderate, severe or none) between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: as for outcome 8
Measure: Number; unit: participants
Groups:
- No Atrophy: Participants with no atrophy at Baseline.
- Mild: Participants with mild atrophy at Baseline.
- Moderate: Participants with moderate atrophy at Baseline.
- Severe: Participants with severe atrophy at Baseline.
Arm/Group | No Atrophy | Mild | Moderate | Severe | No Data
Number analyzed (Participants) | 408 | 57 | 7 | 1 | 33
participants
  Year 5: No atrophy | 306 | 23 | 4 | 1 | 23
  Year 5: Mild atrophy | 7 | 1 | 1 | 0 | 2
  Year 5: Moderate atrophy | 4 | 5 | 1 | 0 | 0
  Year 5: Severe atrophy | 0 | 0 | 0 | 0 | 1
  Year 5: No data | 91 | 28 | 1 | 0 | 7

10. Secondary Outcome: Change From Baseline in Corpus Atrophy
Description: Atrophy was assessed by histopathological examination of cells biopsied from the corpus and classified according to the Sydney classification as mild, moderate, severe or none. The shift table below summarizes the individual transitions in atrophy classification (mild, moderate, severe or none) between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | No Atrophy | Mild | Moderate | Severe | No Data
Number analyzed (Participants) | 451 | 23 | 2 | 0 | 30
participants
  Year 5: No atrophy | 330 | 12 | 1 |  | 17
  Year 5: Mild atrophy | 9 | 0 | 0 |  | 1
  Year 5: Moderate atrophy | 7 | 2 | 1 |  | 0
  Year 5: Severe atrophy | 0 | 1 | 0 |  | 1
  Year 5: No data | 105 | 8 | 0 |  | 11

11. Secondary Outcome: Change From Baseline in Average Antrum Chronic Inflammation Score
Description: Chronic inflammation of the antrum was assessed by histopathology and graded according to the Sydney classification: 0 = None; 1 = mild; 2 = moderate; 3 = Severe
Time Frame: Baseline and Year 5
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole
Number analyzed (Participants) | 506
scores on a scale
  Baseline (n=473) | 0.8 (1.2)
  Change from Baseline (n=353) | -0.2 (1.3)

12. Secondary Outcome: Change From Baseline in Corpus Chronic Inflammation Score
Description: Chronic inflammation of the corpus was assessed by histopathology and graded according to the Sydney classification: 0 = None; 1 = mild; 2 = moderate; 3 = Severe.
Time Frame: Baseline and Year 5
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole
Number analyzed (Participants) | 506
scores on a scale
  Baseline (n=476) | 0.4 (0.8)
  Change from Baseline (n=363) | -0.0 (0.9)

13. Secondary Outcome: Change From Baseline in Antrum Intestinal Metaplasia
Description: Intestinal metaplasia was assessed by biopsy and histopathological examination of the antrum and classified according to the Sydney classification as mild, moderate, severe or none. The shift table below summarizes the individual transitions in intestinal metaplasia classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: as for outcome 8
Measure: Number; unit: participants
Groups:
- None: Participants with no intestinal metaplasia at Baseline.
- Mild: Participants with mild intestinal metaplasia at Baseline.
- Moderate: Participants with moderate intestinal metaplasia at Baseline.
- Severe: Participants with severe intestinal metaplasia at Baseline.
- No Data: Participants with no intestinal metaplasia data at Baseline.
Arm/Group | None | Mild | Moderate | Severe | No Data
Number analyzed (Participants) | 438 | 28 | 7 | 0 | 33
participants
  Year 5: None | 319 | 13 | 4 |  | 23
  Year 5: Mild | 6 | 2 | 2 |  | 2
  Year 5: Moderate | 5 | 1 | 1 |  | 1
  Year 5: Severe | 0 | 0 | 0 |  | 0
  Year 5: No data | 108 | 12 | 0 |  | 7

14. Secondary Outcome: Change From Baseline in Corpus Intestinal Metaplasia
Description: Intestinal metaplasia was assessed by biopsy and histopathological examination of the corpus and classified according to the Sydney classification as mild, moderate, severe or none. The shift table below summarizes the individual transitions in intestinal metaplasia classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | None | Mild | Moderate | Severe | No Data
Number analyzed (Participants) | 472 | 4 | 0 | 0 | 30
participants
  Year 5: None | 359 | 1 |  |  | 18
  Year 5: Mild | 1 | 2 |  |  | 0
  Year 5: Moderate | 0 | 0 |  |  | 1
  Year 5: Severe | 0 | 0 |  |  | 0
  Year 5: No data | 112 | 1 |  |  | 11

15. Secondary Outcome: Change From Baseline in Blood Analysis - Testosterone
Description: The change between testosterone measured at year 5 in males including final visit and Testosterone measured at baseline.
Time Frame: Baseline and Year 5
Population: Safety analysis set, including all male participants who received any study medication. Last observation carried forward was utilized.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Lansoprazole
Number analyzed (Participants) | 285
µg/L
  Baseline (n=285) | 4.57 (1.566)
  Change from Baseline (n=214) | 0.16 (1.275)

16. Secondary Outcome: Change From Baseline in Blood Analysis - Luteinizing Hormone
Description: The change between luteinizing hormone measured at year 5 in males including final visit and luteinizing hormone measured at baseline.
Time Frame: Baseline and Year 5
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Lansoprazole
Number analyzed (Participants) | 286
IU/L
  Baseline (n=286) | 4.73 (3.183)
  Change from Baseline (n=214) | 0.71 (3.101)

17. Secondary Outcome: Change From Baseline in Blood Analysis - Follicle Stimulating Hormone
Description: The change between follicle stimulating hormone (FSH) measured at year 5 in males including final visit and follicle stimulating hormone measured at baseline.
Time Frame: Baseline and Year 5.
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Lansoprazole
Number analyzed (Participants) | 286
IU/L
  Baseline (n=286) | 7.62 (7.864)
  Change from Baseline (n=214) | 0.39 (4.714)

18. Secondary Outcome: Ophthalmologic Examination - Visual Acuity
Description: Visual Acuity was measured using the Snellen eye chart at a distance of 6 meters. Acuity is expressed as a ratio of the test distance (6 M) / the distance the average eye can see the letters on a certain line of the eye chart. Visual acuity of 1 is normal; an individual with acuity of 0.5 could only recognize an object at half the distance compared to an individual with normal acuity.
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lansoprazole
Number analyzed (Participants) | 506
ratio
  Right Eye: Acuity at Baseline (n=443) | 0.927 (0.174)
  Right Eye: Acuity at Year 5 (n=376) | 0.904 (0.186)
  Left Eye: Acuity at Baseline (n=447) | 0.919 (0.181)
  Left Eye: Acuity at Year 5 (n=379) | 0.894 (0.205)

19. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Adaptation Without Glare
Description: Adaptation is the ability of the eye to adjust to various levels of darkness and light. Normal and pathological status of adaptation without glare was defined as follows:
  * Normal status: Contrast between 1:0.05 and 1:23.5.
  * Pathological status: Contrast = 0 or contrast > 1:23.5.
  The shift table below summarizes the individual transitions in the classification of adaptation without glare between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Groups:
- Missing Data: Participants with no data at Baseline.
- Decreased Due to Age: Participants with adaptation decreased due to age at Baseline.
- Pathological: Participants with adaptation classified as pathological at Baseline.
- Normal: Participants with adaptation classified as normal at Baseline.
Arm/Group | Missing Data | Decreased Due to Age | Pathological | Normal
Number analyzed (Participants) | 93 | 7 | 30 | 376
participants
  Year 5: Missing data | 62 | 1 | 4 | 73
  Year 5: Decreased due to age | 0 | 4 | 0 | 1
  Year 5: Pathological | 1 | 0 | 10 | 14
  Year 5: Normal | 30 | 2 | 16 | 288

20. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Adaptation With Glare
Description: Adaptation is the ability of the eye to adjust to various levels of darkness and light. Normal and pathological status of adaptation with glare was defined as follows:
  * Normal status: Contrast between 1:0.05 and 1:23.5.
  * Pathological status: Contrast = 0 or contrast > 1:23.5.
  The shift table below summarizes the individual transitions in the classification of adaptation with glare between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Arm/Group | Missing Data | Decreased Due to Age | Pathological | Normal
Number analyzed (Participants) | 118 | 8 | 52 | 328
participants
  Year 5: Missing data | 75 | 2 | 12 | 58
  Year 5: Decreased due to age | 2 | 4 | 0 | 1
  Year 5: Pathological | 8 | 0 | 16 | 18
  Year 5: Normal | 33 | 2 | 24 | 251

21. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Accommodation
Description: Accommodation is the adjustment of the focal length of the eye lens to keep an object in focus on the retina as its distance from the eye varies, and is measured in diopters: Diopters = 1/(focal length).
Time Frame: Baseline and Year 5
Population: Safety analysis where data were available. Last observation carried forward was utilized.
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Lansoprazole
Number analyzed (Participants) | 506
diopters
  Right Eye: Baseline (n=424) | 2.877 (2.884)
  Right Eye: Change from Baseline (n=348) | -0.090 (2.634)
  Left Eye: Baseline (n=426) | 2.835 (2.831)
  Left Eye: Change from Baseline (n=349) | -0.073 (2.585)

22. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Color Vision
Description: Color vision was assessed by an Ophthalmologist and classified as normal or pathological. Pathological findings include abnormal color vision tests, color blindness and anomalous quotient. Normal indicates no pathological findings were observed. The shift table below summarizes the individual transitions in color vision classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Groups:
- No Data: Participants with no color vision data at Baseline.
- Normal: Participants with normal color vision at Baseline.
- Pathological: Participants with pathological color vision at Baseline.
Arm/Group | No Data | Normal | Pathological
Number analyzed (Participants) | 58 | 406 | 42
participants
  Year 5: No data | 46 | 76 | 5
  Year 5: Normal | 12 | 320 | 10
  Year 5: Pathological | 0 | 10 | 27

23. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Cornea Assessment of Right Eye
Description: The cornea of the right eye was assessed by an Ophthalmologist and judged to be normal or pathological at Baseline and at Year 5. Pathological classification includes abnormal findings such as cataracts, corneal degeneration, opacity, scars or deposits. Normal indicates no pathological findings were observed. The shift table below summarizes the individual transitions in corneal classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Groups:
- Normal: Participants with normal assessment at Baseline.
- Pathological: Participants with pathological assessment at Baseline.
Arm/Group | No Data | Normal | Pathological
Number analyzed (Participants) | 57 | 425 | 24
participants
  Year 5: No data | 46 | 78 | 3
  Year 5: Normal | 11 | 343 | 5
  Year 5: Pathological | 0 | 4 | 16

24. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Cornea Assessment of Left Eye
Description: The cornea of the left eye was assessed by an Ophthalmologist and judged to be normal or pathological at Baseline and at Year 5. Pathological classification includes abnormal findings such as cataracts, corneal degeneration, opacity, scars or deposits. Normal indicates no pathological findings were observed. The shift table below summarizes the individual transitions in corneal classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Arm/Group | No Data | Normal | Pathological
Number analyzed (Participants) | 57 | 429 | 20
participants
  Year 5: No data | 46 | 77 | 4
  Year 5: Normal | 11 | 348 | 5
  Year 5: Pathological | 0 | 4 | 11

25. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Lens Assessment of Right Eye
Description: The lens of the right eye was assessed by an Ophthalmologist and judged to be normal or pathological at Baseline and at Year 5.
  Pathological classification includes abnormal findings such as cataracts, lenticular opacities, vacuoles or pseudophakia. Normal indicates no pathological findings were observed. The shift table below summarizes the individual transitions in lens classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Arm/Group | No Data | Normal | Pathological
Number analyzed (Participants) | 57 | 293 | 156
participants
  Year 5: No data | 46 | 56 | 25
  Year 5: Normal | 8 | 193 | 7
  Year 5: Pathological | 3 | 44 | 124

26. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Lens Assessment of Left Eye
Description: The lens of the left eye was assessed by an Ophthalmologist and judged to be normal or pathological at Baseline and at Year 5.
  Pathological classification includes abnormal findings such as cataracts, lenticular opacities, vacuoles or pseudophakia. Normal indicates no pathological findings were observed. The shift table below summarizes the individual transitions in lens classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Arm/Group | No Data | Normal | Pathological
Number analyzed (Participants) | 57 | 292 | 157
participants
  Year 5: No data | 46 | 56 | 25
  Year 5: Normal | 6 | 193 | 8
  Year 5: Pathological | 5 | 43 | 124

27. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Vitreous Body Assessment of Right Eye
Description: The vitreous body of the right eye was assessed by an Ophthalmologist and judged to be normal or pathological at Baseline and at Year 5.
  Pathological classification includes abnormal findings such as myodesopsia, vitreous opacities, degeneration, detachment or prolapse. Normal indicates no pathological findings were observed. The shift table below summarizes the individual transitions in vitreous body classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Arm/Group | No Data | Normal | Pathological
Number analyzed (Participants) | 57 | 422 | 27
participants
  Year 5: No data | 46 | 73 | 8
  Year 5: Normal | 11 | 338 | 2
  Year 5: Pathological | 0 | 11 | 17

28. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Vitreous Body Assessment of Left Eye
Description: The vitreous body of the left eye was assessed by an Ophthalmologist and judged to be normal or pathological at Baseline and at Year 5.
  Pathological classification includes abnormal findings such as myodesopsia, vitreous opacities, degeneration, detachment or prolapse. Normal indicates no pathological findings were observed. The shift table below summarizes the individual transitions in vitreous body classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Arm/Group | No Data | Normal | Pathological
Number analyzed (Participants) | 59 | 421 | 26
participants
  Year 5: No data | 47 | 73 | 7
  Year 5: Normal | 12 | 341 | 3
  Year 5: Pathological | 0 | 7 | 16

29. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Assessment of Retinal Aspect of the Right Eye
Description: The retinal aspect of the right eye (such as color anomalies) was assessed by an Ophthalmologist and judged to be normal or pathological at Baseline and at Year 5. Pathological classification includes abnormal findings such as deep red ocular fundus, fundus myopicus, retinal disorders, exudates or pigmentation. Normal indicates no pathological findings were observed. The shift table below summarizes the individual transitions in retinal aspect classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Arm/Group | No Data | Normal | Pathological
Number analyzed (Participants) | 59 | 438 | 9
participants
  Year 5: No data | 48 | 80 | 0
  Year 5: Normal | 11 | 356 | 1
  Year 5: Pathological | 0 | 2 | 8

30. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Assessment of Retinal Aspect of the Left Eye
Description: The retinal aspect of the left eye (such as color anomalies) was assessed by an Ophthalmologist and judged to be normal or pathological at Baseline and at Year 5. Pathological classification includes abnormal findings such as deep red ocular fundus, fundus myopicus, retinal disorders, exudates or pigmentation. Normal indicates no pathological findings were observed. The shift table below summarizes the individual transitions in retinal aspect classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Arm/Group | No Data | Normal | Pathological
Number analyzed (Participants) | 57 | 442 | 7
participants
  Year 5: No data | 46 | 80 | 1
  Year 5: Normal | 11 | 361 | 1
  Year 5: Pathological | 0 | 1 | 5

31. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Assessment of Optic Nerve and Papilla of the Right Eye
Description: The optic nerve and papilla of the right eye was assessed by an Ophthalmologist and judged to be normal or pathological at Baseline and at Year 5. Pathological classification includes abnormal findings such as optic nerve cupping, optic nerve cup/disc ratio, or glaucomatous optic disc atrophy. Normal indicates no pathological findings were observed. The shift table below summarizes the individual transitions in optic nerve/papilla classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Arm/Group | No Data | Normal | Pathological
Number analyzed (Participants) | 59 | 422 | 25
participants
  Year 5: No data | 48 | 76 | 4
  Year 5: Normal | 11 | 337 | 4
  Year 5: Pathological | 0 | 9 | 17

32. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Assessment of Optic Nerve and Papilla of the Left Eye
Description: The optic nerve and papilla of the left eye was assessed by an Ophthalmologist and judged to be normal or pathological at Baseline and at Year 5. Pathological classification includes abnormal findings such as optic nerve cupping, optic nerve cup/disc ratio, or glaucomatous optic disc atrophy. Normal indicates no pathological findings were observed. The shift table below summarizes the individual transitions in optic nerve/papilla classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Arm/Group | No Data | Normal | Pathological
Number analyzed (Participants) | 57 | 422 | 27
participants
  Year 5: No data | 46 | 75 | 6
  Year 5: Normal | 11 | 339 | 4
  Year 5: Pathological | 0 | 8 | 17

33. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Assessment of Retinal Blood Vessels of the Right Eye
Description: The retinal blood vessels of the right eye were assessed by an Ophthalmologist and judged to be normal or pathological at Baseline and at Year 5. Pathological classification includes abnormal findings such as retinal vascular disorder, retinopathy, and retinal hemorrhage. Normal indicates no pathological findings were observed. The shift table below summarizes the individual transitions in retinal blood vessel classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Arm/Group | No Data | Normal | Pathological
Number analyzed (Participants) | 59 | 369 | 78
participants
  Year 5: No data | 48 | 68 | 12
  Year 5: Normal | 7 | 279 | 6
  Year 5: Pathological | 4 | 22 | 60

34. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Assessment of Retinal Blood Vessels of the Left Eye
Description: The retinal blood vessels of the left eye were assessed by an Ophthalmologist and judged to be normal or pathological at Baseline and at Year 5. Pathological classification includes abnormal findings such as retinal vascular disorder, retinopathy, and retinal hemorrhage. Normal indicates no pathological findings were observed. The shift table below summarizes the individual transitions in retinal blood vessel classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Arm/Group | No Data | Normal | Pathological
Number analyzed (Participants) | 57 | 369 | 80
participants
  Year 5: No data | 46 | 68 | 13
  Year 5: Normal | 7 | 278 | 7
  Year 5: Pathological | 4 | 23 | 60

35. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Assessment of Macula Lutea of the Right Eye
Description: The macula lutea of the right eye was assessed by an Ophthalmologist and judged to be normal or pathological at Baseline and at Year 5. Pathological classification includes abnormal findings such as maculopathy, retinal pigmentation, macular degeneration, diabetic retinopathy, retinal hemorrhage or aneurysm. Normal indicates no pathological findings were observed. The shift table below summarizes the individual transitions in macula lutea classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Arm/Group | No Data | Normal | Pathological
Number analyzed (Participants) | 60 | 412 | 34
participants
  Year 5: No data | 49 | 75 | 4
  Year 5: Normal | 10 | 317 | 3
  Year 5: Pathological | 1 | 20 | 27

36. Secondary Outcome: Change From Baseline in Ophthalmologic Examination - Assessment of Macula Lutea of the Left Eye
Description: The macula lutea of the left eye was assessed by an Ophthalmologist and judged to be normal or pathological at Baseline and at Year 5. Pathological classification includes abnormal findings such as maculopathy, retinal pigmentation, macular degeneration, diabetic retinopathy, retinal hemorrhage or aneurysm. Normal indicates no pathological findings were observed. The shift table below summarizes the individual transitions in macula lutea classification between Baseline (depicted in the columns) and Year 5 (depicted in the rows).
Time Frame: Baseline and Year 5
Population: Safety analysis set, where data were available. Last observation carried forward was utilized.
Measure: Number; unit: participants
Arm/Group | No Data | Normal | Pathological
Number analyzed (Participants) | 57 | 418 | 31
participants
  Year 5: No data | 46 | 77 | 4
  Year 5: Normal | 10 | 323 | 5
  Year 5: Pathological | 1 | 18 | 22

ADVERSE EVENTS:
Time Frame: Starting with the first administration of study medication for up to 14 days after last dose of study medication.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Lansoprazole
Serious Adverse Events (participants affected / at risk) | 82/506
Other Adverse Events (participants affected / at risk) | 114/506
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lansoprazole (N=506)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 4
Carpal tunnel syndrome (Nervous system disorders) | 1
Restless leg syndrome (Nervous system disorders) | 1
Brain stem infarction (Nervous system disorders) | 1
Carotid sinus syndrome (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Paresis cranial nerve (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Coronary artery disease (Cardiac disorders) | 4
Myocardial infarction (Cardiac disorders) | 3
Atrial flutter (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Pleuropericarditis (Cardiac disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Rectocele (Gastrointestinal disorders) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 2
Concussion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Depression (Psychiatric disorders) | 4
Anxiety disorder (Psychiatric disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Generalised anxiety disorder (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Panic disorder (Psychiatric disorders) | 1
Varicose vein (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Subclavian artery stenosis (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Vascular pseudoaneurysm (Vascular disorders) | 1
Biliary colic (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Neuroborreliosis (Infections and infestations) | 1
Papilloma viral infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Vulval abscess (Infections and infestations) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Chest pain (General disorders) | 1
Impaired healing (General disorders) | 1
Sudden death (General disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Diplopia (Eye disorders) | 1
Toe operation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lansoprazole (N=506)
Bronchitis (Infections and infestations) | 46
Hypertension (Vascular disorders) | 30
Back pain (Musculoskeletal and connective tissue disorders) | 29
Diarrhoea (Gastrointestinal disorders) | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.